CLINICAL TRIAL: NCT00846703
Title: Clinical Study of GD-2008 ALL Protocol for Childhood Acute Lymphoblastic Leukemia in Guangdong Province
Brief Title: The GD-2008 ALL Protocol for Childhood Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Jianpei Fang,MD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007016
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2010-03-08 (Estimated); Status verified 2010-03

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Mercaptopurine; Methotrexate; Vincristine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Protocol A (MM) (Active Comparator)
  Interventions: Drug: 6-mercaptopurine, Methotrexate
- Protocol B (MM/VD) (Experimental)
  Interventions: Drug: 6-mercaptopurine, Methotrexate, Vincristine, Dexamethasone

INTERVENTIONS:
Drug: 6-mercaptopurine, Methotrexate — 6-mercaptopurine p.o. qd
  Methotrexate p.o. qw
  Other Names: For SR and IR patients (Group one)
  Arms: Protocol A (MM)
Drug: 6-mercaptopurine, Methotrexate, Vincristine, Dexamethasone — (1)6-mercaptopurine p.o. qd x 7w Methotrexate p.o. qd x 7w
  (2)Vincristine qw x 1w Dexamethasone p.o. qd x 7d
  Go to (1) and (2)
  Other Names: For SR and IR patients (Group two)
  Arms: Protocol B (MM/VD)

SUMMARY:
The Guangdong work group of childhood acute lymphoblastic leukemia (ALL) therapy was set up in October 2002. The investigators treated the childhood ALL with a GZ2002 protocol since the year 2002, and the protocol was mainly derived from the ALLIC-BFM 2002 protocol. After summarizing the last six years' experience, our group revised the GZ2002 ALL protocol in the year 2008, which is named GD-2008 ALL protocol. The diagnosis and classified criteria is according to the ALLIC-BFM 2002 protocol, and the chemotherapy protocol consists all the therapeutic phases as the ALLIC-BFM 2002 protocol prescribed.

DETAILED DESCRIPTION:
The modification includes:

1. In the induction phase, the agent of dexamethasone 6 mg/m2 is used instead of prednisone after prednisone prophase.
2. The phase "CAM" is 2 weeks for SR patients and 4 weeks for IR and HR patients,respectively.
3. Both the SR and IR treatments involve the protocol mM /M (8 weeks) in the phase of consolidation. However, the folinic acid rescue starts at 36 hours instead of 42 hours. The type of HR enters the block treatment the same with the BFM protocol.
4. There is not randomized study in delayed intensification. The GD-2008 ALL protocol uses the same protocol II with the BFM study.
5. The randomized study focus on the phase of maintenance. The maintenance A is the same with the BFM protocol, while the maintenance B consists of 6mp/MTX and VCR/ dexamethasone. The cycle is 8 weeks: VCR at d1, Dexamethasone at d2 to d7, 6mp from d8 to d56, and MTX at d9,d16, d23, d30, d37,d44,d51.
6. The GD-2008 ALL protocol for HR patients use the re-blocks and protocol II phases.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically proven acute lymphoblastic leukemia (ALL)
* No relapse of a previously unrecognized ALL
* Patients must meet one of the following risk criteria:
* Standard-risk (SR) group meeting all of the following criteria:
* Blasts < 1,000/μL in peripheral blood (PB) on day 8
* Aged 1 to < 6 years
* Initial WBC < 20,000/μL
* M1 (5%) or M2 (≥ 5% to < 25%) blasts in bone marrow on day 15;
* M1 marrow on day 33.
* Intermediate-risk (IR) group meeting all of the following criteria:

  * Aged < 1 or ≥ 6 years and/or WBC ≥ 20,000/μL
  * Blasts < 1,000/μL in PB on day 8
  * M1 or M2 marrow on day 15
  * M3 (≥ 25%) marrow on day 15 OR meets SR criteria but M3 marrow on day 15 and *M1 marrow on day 33.
* High-risk (HR) group meeting ≥ 1 of the following criteria:

  * Meets IR criteria and M3 marrow on day 15 (not SR and M3 on day 15)
  * Blasts ≥ 1,000/μL in PB on day 8
  * M2 or M3 marrow on day 33
  * Translocation t(9;22) [BCR/ABL+] (Philadelphia chromosome-positive) or t(4;11) [MLL/AF4+].

Exclusion Criteria:

* No Down syndrome
* No other major disease that prohibits study treatment (e.g., severe congenital heart disease)
* Not requiring significant therapy modification owing to study therapy associated complications
* No complications due to other interventions
* No one with missing data that are needed for the differential diagnosis, or for selection of the proper therapy arm

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2008-07; Primary Completion 2013-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The improvement of safety in the treatment protocol | Two months

CONTACTS AND LOCATIONS:
Overall Officials: Jianpei Fang, M.D., Study Director — Second Affiliated Hospital, Sun Yat-Sen University; Xuequn Luo, M.D., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University; Jianliang Chen, M.D., Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University; Xiaofei Sun, Principal Investigator — The cancer hospital of Sun Yat-sen University; Xuedong Wu, Principal Investigator — Nanfang hospital of Nanfang Medical University; Liming Tu, M.D., Principal Investigator — Guangdong Provincial People's Hospital; Dongbo Lai, M.D., Principal Investigator — Guangzhou children's hospital; Changgang Li, M.D., Principal Investigator — Shenzhen Children's Hospital; Liyang Liu, M.D., Principal Investigator — Huizhou People's Central Hospital
Locations (1):
- The second affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China